CLINICAL TRIAL: NCT07183007
Title: Development of a Dietary Intervention Model Based on Genetic Data as an Implementation of a Healthy Lifestyle in the Management of Systemic Lupus Erythematosus Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Alvina Widhani, Sp.PD, KAI, Associate Professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KET948/UN2F1/ETIK/PPM0002/2025
Record Dates: First submitted 2025-08-28; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; dietary intervention; nutrigenomic; HLA-DQ2; HLA-DQ8
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention based on genetic data (Active Comparator): Dietary intervention with low gluten diet for systemic lupus patients with HLA-DQ2 or HLA-DQ8 positive
  Interventions: Other: Low gluten diet
- Control group (No Intervention): Usual diet for systemic lupus erythematosus patients with HLA-DQ2 or DQ8 positive

INTERVENTIONS:
Other: Low gluten diet — Systemic lupus erythematosus patients with HLA-DQ2 or DQ-8 positive will be randomized to dietary intervention group or control group. Those who are randomized to dietary intervention group will get dietary planning and intervention from a nutritionist with low gluten diet
  Arms: Dietary intervention based on genetic data

SUMMARY:
The goal of this clinical trial is to learn if dietary intervention based on genetic data benefits in the management of systemic lupus erythematosus patients. It will also learn about the safety of this intervention. The main questions it aims to answer are:

* What is the effect of dietary intervention based on genetic data as part of a healthy lifestyle in the management of SLE patients on disease activity?
* What is the effect of dietary intervention based on genetic data as part of a healthy lifestyle in the management of SLE patients on quality of life Researchers would compare dietary intervention based on genetic data to a no intervention to see if dietary intervention based on genetic data improves disease activity and quality of life of SLE patients.

Participants will:

* Be checked for genetic test (HLA DQ2 and DQ8) as screening
* Be randomized to dietary intervention group or control group if has HLA DQ2 or DQ8 positive from screening
* Visit the clinic once every month for checkups and lab test if were randomized to dietary intervention group or control group
* Do food record as instructed if were randomized to dietary intervention group or control group

ELIGIBILITY:
Inclusion Criteria:

1. Patients with systemic lupus erythematosus (SLE) diagnosed according to the 2019 EULAR/ACR criteria, registered as patients at RSCM.
2. Age above 18 years

Exclusion Criteria:

1. Presence of active infection.
2. Refusal to participate in the study.
3. Pregnancy.
4. Breastfeeding.
5. Already on a specific autoimmune-related diet.
6. Patients with severe medical conditions (active cancer, stage V chronic kidney disease, or acute heart failure).
7. Patients taking corticosteroids equivalent to more than 20 mg/dL prednisone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-21 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Systemic Lupus Erythematosus (SLE) Disease Activity | baseline, 1 month after intervention and 3 months after intervention
  Measurement of Systemic Lupus Erythematosus disease activity using The Mexican Systemic Lupus Erythematosus Disease Activity Index (MEX SLEDAI). Minimal score is 0 and maximal score is 32. Score 0-1 indicate remission; 2-5 indicate mild disease activity; 6-9 indicate moderate disease activity; 10-13 indicate severe disease activity; and ≥14 indicate very severe disease activity
Lupus Quality of life | baseline, 1 month after intervention and 3 months after intervention
  Measurement of the Quality of Life (QOL) of Systemic Lupus Erythematosus patient using the LupusQOL, a disease-specific, 34-item instrument that assesses eight domains: physical health pain, planning, intimate relationship, emotional health, burden to others, body image, and fatigue. Each item uses a 5-point Likert scale (0-4), with domain scores calculated by averaging item responses within each domain, dividing by four, and multiplying by 100 to yield scores ranging from 0 (worst) to 100 (best QoL)

SECONDARY OUTCOMES:
Fatigue score | baseline, 1 month after intervention, and 3 months after intervention
  Fatigue score is measured using the Fatigue Severity Scale, a 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity according to a self-report scale. The items are scored on a 7-point scale with 1 = strongly disagree and 7= strongly agree.
  The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
Physical activity | baseline, 1 month after intervention, and 3 months after intervention
  Measuring physical activity using short form of International Physical Activity Questionnaire. This questionnaire provides information on the time spent walking, in vigorous- and moderate intensity activity and in sedentary activity in the last 7 days to estimate total physical activity in MET-min/week and time spent sitting
Sleep quality | baseline, 1 month after intervention, and 3 months after intervention
  Measuring sleep quality using Pittsburgh Sleep Quality Index (PSQI). It differentiates "poor" from "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale.
  A global sum of "5" or greater indicates a "poor" sleeper. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Anxiety and depression | baseline, 1 month after intervention, and 3 months after intervention
  Measuring anxiety and depression score using Hospital Anxiety Depression Scale (HADS). The HADS is a 14-item questionnaire consists of two subscales: one for anxiety (HADS-A) and one for depression (HADS-D), each containing 7 items. Respondents rate their feelings over the past week on a 4-point Likert scale, where: 0 = Not at all; 1 = Occasionally; 2 = Often; 3 = Most of the time. The total score can range from 0 to 42, combining both anxiety and depression scores. Each subscale (anxiety and depression) can score between 0 and 21.
  Interpretation of Scores: 0-7= Normal; 8-10: Mild symptoms; 11-21: Moderate to severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because it is not included in the informed consent

REFERENCES:
- [Derived] Widhani A, Wardhani WI, Shahab SN, Kasih M, Cahyanur R, Yunihastuti E, Ahani AR. Dietary Intervention for Systemic Lupus Erythematosus patients based on HLA-DQ2 and DQ8 genotyping (DISH): a protocol for a randomised controlled study. Lupus Sci Med. 2025 Nov 24;12(2):e001833. doi: 10.1136/lupus-2025-001833. PMID 41290265